CLINICAL TRIAL: NCT04610749
Title: Diabetic Retinopathy as a Marker of Cognitive Dysfunction and Depression
Acronym: DIRMA
Status: Completed | Type: Observational
Sponsor: Region of Southern Denmark (Other)
Responsible Party: Principal Investigator, Frederik Nørregaard Pedersen, Principal Investigator, Region of Southern Denmark
Other Study IDs: S-20200050
Record Dates: First submitted 2020-10-22; First posted 2020-10-30 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-04

CONDITIONS: Diabetic Retinopathy; Depression; Cognitive Impairment; Cognitive Dysfunction
MeSH Terms: conditions — Diabetic Retinopathy; Depression; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In recent years damage to the nerve fibers in the retina has been experienced as an early sign of complications resulting from type 2 diabetes.

In addition, it has been presented that people with type 2 diabetes are at increased risk of developing brain diseases, such as mild memory impairment and Alzheimer's disease, as well as mental illness in the form of depression.

The eye corresponds to be a protruding part of the brain which means the brain and the eye share common features.

Currently it is time and cost consuming to asses changes in the brain, but recent research has shown that patient friendly eye examinations can detect nerve loss brain diseases.

Recent studies have shown that depression can also have a physiological component, which can be measured by changes in structures in the retina of the eye.

In this research project, we will conduct a clinical study, to assess whether there is an association between changes in the retina of the eye (e.g. vascular structure, retinal thickness and oxygen saturation) and mild memory impairment and depression respectively in people with type 2 diabetes.

The clinical study will help to clarify the possibility of including patient-friendly eye examinations in the assessment of minimal memory impairment and depression in patients with type 2 diabetes.

200 people with type 2 diabetes will be invited to participate in a clinical cross-sectional study. The Funen Diabetes Database will be used as recruitment tool. Participants will undergo a thorough eye examination as well as neuropsychological examinations for signs of mild memory impairment. They will also complete questionnaires regarding depressive symptoms.

Overall, the research project will help to create awareness in this area among both healthcare professionals and patients. Early risk detection could mean better diabetes care and fewer complications, which will have a major impact on quality of life and contribute to socio-economic gains. Any findings may contribute to the discussion of individualized screening and treatment if some individuals within this group are at increased risk of developing memory impairment or depression.

DETAILED DESCRIPTION:
A cross sectional study will be performed to determine correlation between retinal endpoints in persons with type 2 diabetes and cognitive impairment. 200 patients with type 2 diabetes without diabetic retinopathy and non to severe diabetic retinopathy.

Primary objective:

To determine whether structural and/or metabolic retinal markers are able to differentiate people with minimal cognitive impairment (MCI) within persons with type 2 diabetes (T2D).

Secondary objective

1. To assess whether retinal metabolism measured by oximetry can identify individuals with MCI among people with T2D.
2. To assess whether retinal metabolism measured by oximetry can identify individuals with depressive symptoms among people with T2D.
3. To determine whether retinal structural markers can identify people with depressive symptoms among people with T2D.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes
2. 65 years and older
3. Diabetes duration of at least 5 years
4. None to severe non-proliferative DR (NPDR), as determined by the evaluating ophthalmologists using fundus examination by slit-lamp biomicroscopy or fundus imaging.
5. Able to provide informed consent

Exclusion Criteria:

1. Previous history of stroke or neurodegenerative diseases.
2. Proliferative DR (PDR), Diabetic Macular Edema (DME) or other eye disorders affecting vision besides these complications of DR.
3. Previous laser photocoagulation.
4. Other diseases which may induce retinal neurodegeneration (e.g. glaucoma).
5. Subjects with a refractive error ≥ ± 6 D.
6. Media opacities that preclude retinal imaging.
7. Severe systemic illness or personal circumstances that would not make it possible for the patients to fulfil study protocols.

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: Patients with type 2 diabetes
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2020-11-25 (Actual); Primary Completion 2022-02-25 (Actual); Study Completion 2022-02-25 (Actual)

PRIMARY OUTCOMES:
Retinal metabolism | 1 day
  Measured by retinal oximetry

SECONDARY OUTCOMES:
Retinal neurodegeneration | 1 day
  Measured by Spectral Domain Optical Coherence Tomography
Central Retinal vascular abnormalities | 1 day
  Measured by fundus photography and analyzed with semi automated software
Retinal vascular abnormalities | 1 day
  Measured by Optical Coherence Tomography Angiography
Depressive symptoms | 1 day
  Measured by Geriatric depression scale GDS-15 and Measured by Inventory of depressive symptomatology (Self-report)

CONTACTS AND LOCATIONS:
Overall Officials: Frederik N Pedersen, M.D, Principal Investigator — Department of Ophthalmology, OUH
Locations (1):
- Odense University Hospital, Odense, Fyn, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
•Undecided: It is not yet known if there will be a plan to make IPD available